CLINICAL TRIAL: NCT06595511
Title: Development of a Sensory Entrainment-Integrated Cognitive Game Kit to Improve Cognitive Functions in Alzheimer's Disease
Brief Title: Effects of Combined 40 Hz Audio-visual Stimulation and Cognitive Games on Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other); Guven Health Group (Other)
Responsible Party: Principal Investigator, Bahar Güntekin, Prof. Dr., Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-6692
Record Dates: First submitted 2024-08-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer's Disease; 40 Hz Stimulation; EEG Brain Oscillations
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Alzheimer's Disease Treatment Group (Active Comparator): The group will engage with the 40 Hz sensory entrainment-integrated cognitive game kit for one hour a day, five days a week, for three months.
  Interventions: Device: Sensory Entrainment-Integrated Cognitive Game Kit
- Alzheimer's Disease Control Group (No Intervention)
- Healthy Older Adult Group (No Intervention)

INTERVENTIONS:
Device: Sensory Entrainment-Integrated Cognitive Game Kit — Active comparator group will engage with the 40 Hz sensory entrainment-integrated cognitive game kit for one hour a day, at least five days a week, for three months.
  Arms: Alzheimer's Disease Treatment Group

SUMMARY:
In addition to ongoing drug treatments for Alzheimer Disease (AD), protective approaches that can halt the progression of the disease are of particular importance. This project aims to develop a digital application that can monitor cognitive impairment, using EEG findings proven effective at the clinical level in Alzheimer and various types of dementia, including sensory entrainment and digital cognitive games.

To this end, a collaboration between Istanbul Medipol University and Güven Future Health Technologies Inc. will develop a device featuring audio-visual sensory entrainment and digital cognitive games. This device will be made available to Alzheimer patients, and the differences between patients who use the application for three months, patients who do not use the application, and healthy controls will be evaluated through neurological examinations, neuropsychological tests, and EEG recordings indicating cognitive functions by the neurologist, project coordinator, and bursars. Monthly assessments, including EEG recordings, will also continue at home, and an application will be created to evaluate changes in cognitive functions through EEG data.

By the end of the project, an application that includes sensory entrainment and digital cognitive games, proven effective at the clinical level using EEG findings for Alzheimer dementia patients, will be developed. Additionally, a health kit capable of temporal monitoring of cognitive function changes through EEG data will have been developed.

DETAILED DESCRIPTION:
This study aims to recruit early and middle-stage Alzheimer patients aged between 60 and 75, along with age and gender-matched healthy older adults. Two different Alzheimer groups will be created: one group will utilize a 40 Hz sensory entrainment-integrated cognitive game kit at home, while the other group will not receive any treatment. The treatment group will comprise 10 Alzheimer patients who will engage with the 40 Hz sensory entrainment-integrated cognitive game kit for 1 hour a day, at least five days a week, for three months. Comprehensive neuropsychological assessments and electroencephalography (EEG) recordings will be conducted in the laboratory on the first day, followed by mobile EEG recordings at home at the end of the first and second months. After three months of using the sensory entrainment/cognitive game kit, the participants will again undergo neuropsychological assessment and EEG recording in the laboratory. The second Alzheimer group (n=10) will not be administered any treatment and will undergo the same assessment protocol as the treatment group. Furthermore, in addition to these two groups, a healthy older adult group (n=10) will also be included in the study, with assessments scheduled only on the first day and at the end of the third month.

ELIGIBILITY:
Inclusion and Exclusion Criteria for Alzheimer Patients:

Inclusion Criteria:

* Diagnosed with AD according to DSM-IV and NINCDS-ADRDA criteria,
* Impaired activities of daily living,
* Having a CDR score of 1-2 and an SMMT score of 15-26,
* Stable use of psychoactive medications, including acetylcholinesterase inhibitors or other medications that enhance cognitive functions,
* Individuals aged 60-86 with at least 5 years of education.

Exclusion Criteria:

* Having frontotemporal dementia, vascular dementia, Lewy body dementia or other types of dementia,
* Parkinsonism, clinical depression, other mental disorders, epilepsy, drug addiction, alcohol addiction, and traumatic brain injury

Inclusion and Exclusion Criteria of Healthy Older Adults:

Inclusion criteria:

* Between the ages of 60-86
* Without any neurological abnormalities or general cognitive impairment (MMSE above 25),
* Not diagnosed with a neurological and/or psychiatric disease,
* Not using neurological and/or psychiatric medication

Exclusion criteria

* Having clinical signs of cognitive impairment, such as mild cognitive impairment, Alzheimer disease, Parkinson disease, Lewy body dementia, frontotemporal dementia, etc.
* Epilepsy, alcohol and/or drug addiction, use of medications that affect cognitive functions, and traumatic brain injury

Ages: 60 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
EEG recording | At baseline and month 3
  EEG will be recorded under these conditions:
  * Spontaneous EEG (8 minutes eyes open, 8 minutes eyes closed)
  * Visual oddball
  * Auditory oddball
  * 40 Hz flicker stimulation EEG recording (8 minutes eyes open, 8 minutes eyes closed)

SECONDARY OUTCOMES:
Standardized Mini Mental State Examination (SMMSE) | At baseline and month 3
  For the comprehensive cognitive status
Verbal memory processes test (Öktem-SBST) and Wechsler Visual Production Subtest | At baseline and month 3
  For the assessment of memory functions
WMS-R Digit Span Test | At baseline and month 3
  For the assessment of attention
Stroop Test, Clock Drawing Test, Verbal Fluency Tests (categorical and phonemic) and Trail Making Test | At baseline and month 3
  For the assessments of executive function
Boston Naming Test | At baseline and month 3
  For the assessment of language functions
Benton Line Orientation Test and Benton Face Recognition Test | At baseline and month 3
  For the assessment of visuospatial functions

OTHER OUTCOMES:
Mobile EEG recording at home | month 1 and 2
  EEG will be recorded under these conditions:
  * Spontaneous EEG (8 minutes eyes open, 8 minutes eyes closed)
  * 40 Hz flicker stimulation EEG recording (8 minutes eyes open, 8 minutes eyes closed) Delta, theta, alpha, beta, gamma power spectrum and phase locking indexes will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided